CLINICAL TRIAL: NCT00121238
Title: Phase II Evaluation of EMD 121974 (NSC 707544, Cilengitide) in Patients With Non-Metastatic Androgen Independent Prostate Cancer
Brief Title: Cilengitide in Treating Patients With Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03066; 2004-045 (Other: University of Michigan Comprehensive Cancer Center); N01CM62206 (NIH); CDR0000438708 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2005-07-19; First posted 2005-07-21 (Estimated); Results first posted 2016-04-28 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2013-02

CONDITIONS: Recurrent Prostate Cancer; Stage I Prostate Cancer; Stage IIA Prostate Cancer; Stage IIB Prostate Cancer; Stage III Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Cilengitide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental treatment: cilengitide (Experimental): Patients receive cilengitide IV over 1 hour on days 1, 4, 8, 11, 15, 18, 22, and 25. Treatment repeats every 28 days for at least 3 courses in the absence of disease progression or unacceptable toxicity. After 3 courses, patients undergo evaluation. Patients achieving a complete prostate-specific antigen (PSA) response (i.e., PSA < 0.2 ng/mL) receive 2-3 additional courses of therapy. Patients with partial PSA response or stable disease continue treatment indefinitely in the absence of disease progression or unacceptable toxicity. Patients demonstrating disease progression by CT scan, MRI, or bone scan are removed from the study.
  Interventions: Drug: cilengitide

INTERVENTIONS:
Drug: cilengitide — Given IV
  Other Names: EMD 121974

SUMMARY:
This phase II trial is studying how well cilengitide works in treating patients with prostate cancer. Cilengitide may stop the growth of prostate cancer by blocking blood flow to the tumor

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the rate of Prostate Specific Antigen response associated with EMD121974 therapy in patients with non-metastatic androgen-independent prostate cancer.

SECONDARY OBJECTIVES:

I. To evaluate the safety of EMD121974 in patients with non-metastatic androgen-independent prostate cancer.

II. To assess the change in the slope of Prostate Specific Antigen associated with EMD121974 in patients with non-metastatic androgen-independent prostate cancer.

III. To assess response duration, time to progression and survival.

TERTIARY OBJECTIVES:

I. To determine the effects of integrin αvβ3 and αvβ5 inhibition on total circulating tumor and endothelial cells isolated from peripheral blood and bone marrow aspirates from patients with non-metastatic androgen-independent prostate cancer.

II. To study the genotypic/phenotypic variances in circulating tumor cells in patients with non-metastatic androgen-independent prostate cancer before and after EMD121974 treatment.

III. To develop a genetic profile by cDNA microarray analysis of circulating tumor cells isolated from patients with non-metastatic androgen-independent prostate cancer before and after integrin αvβ3 and αvβ5 inhibition.

OUTLINE: This is an open-label, multicenter study.

Patients receive cilengitide IV over 1 hour on days 1, 4, 8, 11, 15, 18, 22, and 25. Treatment repeats every 28 days for at least 3 courses in the absence of disease progression or unacceptable toxicity. After 3 courses, patients undergo evaluation. Patients achieving a complete prostate-specific antigen (PSA) response (i.e., PSA < 0.2 ng/mL) receive 2-3 additional courses of therapy. Patients with partial PSA response or stable disease continue treatment indefinitely in the absence of disease progression or unacceptable toxicity. Patients demonstrating disease progression by CT scan, MRI, or bone scan are removed from the study.

ELIGIBILITY:
Inclusion Criteria:

* A histologic or cytologic diagnosis of prostate cancer
* No evidence of metastatic disease, or local progression
* PSA-only progression despite androgen deprivation therapy and antiandrogen withdrawal (28 days for flutamide and 42 days for bicalutamide or nilutamide); PSA progression is defined as 3 consecutive rising levels, with an interval of > 1 week between each determination; the last determination must have a minimum value of >= 2 ng/ml and be determined within two weeks prior to registration

  * If the third confirmatory value is less than the previous value, the patient will still be eligible if a repeat value (No. 4) is found to be greater than the second value
* Patients must continue on LHRH agonists; they also may continue on any stable doses (considered stable, if on current medicine dosing for one month or longer) of megace or corticosteroids; they must be off all other therapies intended to treat the cancer for 4 weeks
* ECOG performance status of 0-2
* No prior EMD 121974 therapy is allowed
* No investigational or commercial agents or therapies may be administered with the intent to treat the patient's malignancy
* Testosterone < 50 ng/dl; patients must continue primary androgen deprivation with an LHRH agonist, if they have not undergone orchiectomy
* Four weeks must have elapsed since major surgery
* Life expectancy of greater than 6 months
* Patients must have normal organ and marrow function as defined below obtained within 14 days prior to registration:
* ANC >= 1,500/µl
* Platelet count >= 100,000/ µl
* Creatinine =< 1.5 x upper limits of normal
* Bilirubin within normal limits
* SGOT (AST) =< 2.5 x upper limits of normal
* SGPT (ALT) =< 2.5 x upper limits of normal
* PSA >= 2 ng/ml
* The effects of EMD 121974 on the developing human fetus at the recommended therapeutic dose are unknown; for this reason and because antiangiogenic agents are known to be teratogenic, men must agree to use adequate contraception prior to study entry and for the duration of study participation
* Ability to understand and the willingness to sign a written informed consent that is approved by the Institutional Human Investigation Committee

Exclusion Criteria:

* Patients may continue on a daily Multi-Vitamin, but all other herbal, alternative and food supplements (i.e. PC-Spes, Saw Palmetto, St John Wort, etc.) must be discontinued before registration
* Patients on stable doses of bisphosphonates which have been started no less than 6 weeks prior to protocol therapy, that show subsequent PSA progression, may continue on this medication, however patients are not allowed to initiate bisphosphonate therapy immediately prior or during the study
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients with a "currently active" second malignancy, other than non-melanoma skin cancers or superficial bladder cancer, are not eligible; patients are not considered to have a "currently active" malignancy if they have completed therapy and are now considered without evidence of disease for 2 years

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2005-01; Primary Completion 2010-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maha Hussain, Principal Investigator — University of Michigan University Hospital
Locations (1):
- University of Michigan University Hospital, Ann Arbor, Michigan, United States

REFERENCES:
- [Result] Alva A, Slovin S, Daignault S, Carducci M, Dipaola R, Pienta K, Agus D, Cooney K, Chen A, Smith DC, Hussain M. Phase II study of cilengitide (EMD 121974, NSC 707544) in patients with non-metastatic castration resistant prostate cancer, NCI-6735. A study by the DOD/PCF prostate cancer clinical trials consortium. Invest New Drugs. 2012 Apr;30(2):749-57. doi: 10.1007/s10637-010-9573-5. Epub 2010 Nov 4. PMID 21049281

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 16 patients were registered to the protocol at 6 centers between January 2005 and May 2007.
Pre-assignment Details: 1 patient progressed clinically before any treatment and was not included in toxicity or efficacy endpoint analysis. Two patients who received drug were deemed ineligible because of PSA rise requirement and withdrawn for analysis for efficacy but their data was entered into toxicity analysis
Groups:
- Drug Treatment (Cilengitide): Patients receive cilengitide IV over 1 hour on days 1, 4, 8, 11, 15, 18, 22, and 25. Treatment repeats every 28 days for at least 3 courses in the absence of disease progression or unacceptable toxicity. After 3 courses, patients undergo evaluation. Patients achieving a complete prostate-specific antigen (PSA) response (i.e., PSA < 0.2 ng/mL) receive 2-3 additional courses of therapy. Patients with partial PSA response or stable disease continue treatment indefinitely in the absence of disease progression or unacceptable toxicity. Patients demonstrating disease progression by CT scan, MRI, or bone scan are removed from the study.
  cilengitide : Given IV
  Experimental drug treatment : Correlative studies
Period: Overall Study
Arm/Group | Drug Treatment (Cilengitide)
Started | 16
Completed | 13 (2 were later deemed ineligible (PSA rise), censored from efficacy but included for toxicity analysis)
Not Completed | 3
Not completed — disease progression before intervention | 1
Not completed — Protocol Violation | 2

BASELINE CHARACTERISTICS:
Population: 16 patients were enrolled but only 13 were analyzed. 1 patient progressed clinically before any treatment.Two patients who received study drug were deemed ineligible as they did not meet entry PSA criteria of three consecutive rises in PSA.
Arm/Group | Drug Treatment (Cilengitide)
Number analyzed (Participants) | 13
Age, Customized [Median (Full Range); unit: years]
  age in years | 65.5 [53.8 to 78.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 13
Prostate Specific Antigen (PSA) [Median (Full Range); unit: ng/mL] | 8.4 [2.2 to 77]
Gleason sum [Number; unit: participants] — A Gleason score is given to prostate cancer based upon its microscopic appearance. Gleason scores range from 2 to 10, with 2 representing the most well-differentiated tumors (more favorable prognosis) and 10 the least-differentiated tumors (less favorable prognosis).
  participants
    Gleason sum 6 | 2
    Gleason sum 7 | 6
    Gleason sum 8 | 2
    Gleason sum 9 | 3
Karnofsky Performance Score [Median (Full Range); unit: units on a scale] — A standard way of measuring the ability of cancer patients to perform ordinary tasks. The Karnofsky performance scores range from 0- 100. A higher score means the patient/participant is better able to conduct daily activities.
  units on a scale | 90 [80 to 100]
Prior radiation to prostate [Number; unit: participants] — Of the 13 patients analyzed, only 11 patients had prior radiation.
  participants
    Definitive | 5
    Adjuvant | 3
    Salvage | 3
Radical Prostatectomy [Number; unit: participants] — Surgery to manage prostate cancer by removal of the patient's prostate and vesicles.
  participants | 6
No Local Treatment Modality [Number; unit: participants] — 2 of the 13 patients analyzed had no local treatment modality.
  participants | 2
Median time since ADT initiation [Median (Full Range); unit: years] — Median time after initiation of Androgen Deprivation Treatment (ADT)
  years | 4.7 [1 to 10.6]

OUTCOME MEASURES:

1. Primary Outcome: The Number of Patients With a PSA Decline of ≥50%
Description: To assess the rate of Prostate Specific Antigen response associated with EMD121974 therapy in patients with non-metastatic androgen-independent prostate cancer.
  This measure defined as a drop in PSA of at least 50% from the final pre-treatment value.
Time Frame: Up to 5 years
Population: Per protocol: of the 16 patients registered for this arm, 13 were analyzed. 1 patient lost eligibility due to disease progression, 2 others were censored from efficacy analysis because it was determined they were ineligible based on PSA requirements.
Measure: Number; unit: participants
Arm/Group | Drug Treatment (Cilengitide)
Number analyzed (Participants) | 13
participants | 0

2. Secondary Outcome: Median PSA Slope Difference
Description: Median PSA slope difference was calculated between baseline and 6 months.
Time Frame: Baseline to 6 months
Measure: Median (Inter-Quartile Range); unit: ng/mL/month
Arm/Group | Drug Treatment (Cilengitide)
Number analyzed (Participants) | 13
ng/mL/month | 0.9 [-0.97 to 4.11]
Statistical Analysis 1: Comparison: Drug Treatment (Cilengitide); Test type: Superiority or Other; p = 0.27, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: The Number of Participants With at Least One Incident of Toxicity
Description: Toxicity was evaluated by NCI-CTCAE (ver. 3) criteria in all 15 treated patients (16 patients were enrolled however one progressed prior to treatment) including the two ineligible patients.
Time Frame: Up to 5 years
Population: All treated patients, including 2 patients who were deemed ineligible for the study's endpoints to measure efficacy.
Measure: Number; unit: participants
Arm/Group | Drug Treatment (Cilengitide)
Number analyzed (Participants) | 15
participants | 15

4. Secondary Outcome: Median Survival Time
Description: 6 of 13 patients were alive at five years. The Median survival time was calculated for all patients.
Time Frame: Up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Drug Treatment (Cilengitide)
Number analyzed (Participants) | 13
months | 34.5 [27.4 to NA] — The upper limit has not yet been reached.

5. Secondary Outcome: Mean Time to Progression of Prostate Cancer
Description: Kaplan-Meier estimates of time to progression will be reported.
Time Frame: Up to 5 years
Population: Patients were eligible if they had a histologic or cytologic diagnosis of prostate cancer with no evidence of metastatic disease or local progression on radiologic imaging and had 3 consecutive rising levels of prostate specific antigen (psa). Eligible patients who were treated on this trial were analyzed for survival
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | Drug Treatment (Cilengitide)
Number analyzed (Participants) | 13
months | 1.8 [0.9 to 2.8]

ADVERSE EVENTS:
Time Frame: During treatment with study drug for 1 year if toxicity did not halt treatment
Description: Toxicity was evaluated by NCI-CTCAE (ver. 3) criteria in all 15 treated patients including the 2 ineligible patients. No Grade 4 events,2 grade 3 events, 3 grade 2 events and 22 grade 1 adverse events.
Arm/Group | Drug Treatment (Cilengitide)
Serious Adverse Events (participants affected / at risk) | 2/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Drug Treatment (Cilengitide) (N=15)
atrial fibrillation (Cardiac disorders) | 2 — 2 CTCAE Grade 3 atrial fibrillation occured in 2 separate patients
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Drug Treatment (Cilengitide) (N=15)
Arthritis (Gr1) (Musculoskeletal and connective tissue disorders) | 2 — 2 events of Gr1 arthritis
Increased aspartate aminotransferase (Gr1) (Blood and lymphatic system disorders) | 1 — Gr1 event affecting 1 patient
Constipation (Gr1) (Gastrointestinal disorders) | 1 — 1 occurence of Gr1 constipation
Diarrhea (Gr1) (Gastrointestinal disorders) | 1 — 1 occurrence of Gr1 diarrhea
Dry eye syndrome (Gr1) (Eye disorders) | 1 — 1 occurence of grade 1 dry eye syndrome
Edema (Gr.1) (General disorders) | 1 — 1 occurence of Gr. 1 edema
Fatigue (Gr.1) (General disorders) | 4 — 4 occurences of Gr.1 fatigue
Flushing (Gr1) (General disorders) | 1 — 1 occurence of Gr.1 flushing
Headache (Gr.1) (General disorders) | 1 — One occurrence of Gr1 headache
Decreased hemoglobin (gr1) (Blood and lymphatic system disorders) | 2 — 2 occurences of decreased hemoglobin
Hyperglycemia NOS (Gr.1) (Metabolism and nutrition disorders) | 1 — 1 instance of Gr1 Hyperglycemia
Hyperglycemia (Gr.1) (Metabolism and nutrition disorders) | 1 — 1 instance of Gr1 Hyperglycemia
Hyponatremia (Gr.1) (General disorders) | 1 — 1 instance of gr.1 hyponatremia
Memory impairment (Gr.1) (Nervous system disorders) | 1 — 1 instance of Gr.1 memory impairment
Nausea Gr 1 (Gastrointestinal disorders) | 1 — 1 instance of Gr.1 nausea
Rash (desquamating) (Gr.1) (Skin and subcutaneous tissue disorders) | 1 — 1 instance of grade 1 rash
Toothache (Gr.1) (Gastrointestinal disorders) | 1 — 1 instance of grade 1 toothache
Dyspnea (Gr.2) (Respiratory, thoracic and mediastinal disorders) | 1 — 1 instance of grade 2 dyspnea
Lymphopenia (Gr.2) (Blood and lymphatic system disorders) | 1 — 1 incident of grade 2 lymphopenia
Osteonecrosis (Gr.2) (Musculoskeletal and connective tissue disorders) | 1 — 1 instance of grade 2 osteonecrosis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less